CLINICAL TRIAL: NCT05453201
Title: Developing an Integrative, Recovery-Based, Post-Acute COVID-19 Syndrome (PACS) Psychotherapeutic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4092-P; 1I21RX004092-01A1 (NIH)
Record Dates: First submitted 2022-07-05; First posted 2022-07-12 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
Keywords: COVID-19; Functional Improvement; Long-Haul COVID; Mental Health; Post-Acute COVID-19 Syndrome (PACS)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Psychological Well-Being | interventions — Salvage Therapy; Methods

STUDY DESIGN:
Intervention Model Description: PACS Patients will be recruited through recruitment from James J. Peters VAMC PACS clinical program and clinician referrals. The Bronx had significantly higher rates of COVID-19 infection than other boroughs in New York City. Thus, recruitment of up to 36 Veterans is feasible within the 18-month timeframe.
  Veterans will participate in a LCCR group (1x/week for a total of 16 sessions) via the HIPAA-compliant telehealth platform VA Video Connect (VVC) and/or VA WebEx with two co-therapists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long COVID Coping and Recovery (LCCR) Intervention (Experimental): Veterans will participate in a LCCR (1x/week for a total of 16 sessions) via the HIPAA-compliant telehealth platform VA Video Connect (VVC) and/or VA WebEx with two co-therapists.
  Interventions: Behavioral: Long COVID Coping and Recovery (LCCR) Intervention

INTERVENTIONS:
Behavioral: Long COVID Coping and Recovery (LCCR) Intervention — Veterans will participate in a LCCR (1x/week for a total of 16 sessions) via the HIPAA-compliant telehealth platform VA Video Connect (VVC) and/or VA WebEx with two co-therapists.

SUMMARY:
Post-Acute COVID-19 Syndrome (PACS), colloquially known as Long COVID, is a prevalent phenomenon that affects thousands of Veterans in VA care. VA patients suffering from Long COVID not only experience lingering physical symptoms following COVID-19 infection, but have increased mental health problems including sleep disorders, anxiety disorders, trauma and stress-related disorders as well as increased use of opioid and non-opioid pain medications, antidepressants, and sedatives to treat these conditions. Developing recovery-oriented care, "a process of change through which individuals improve their health and wellness, live a self-directed life, and strive to reach their full potential" is a VA priority, however available Long COVID treatments primarily target symptom relief and are not designed to promote the recovery and rehabilitation of Veterans in a mental health context. Long COVID Coping and Recovery (LCCR) is a promising manualized, recovery-focused psychotherapeutic group intervention which aims to improve psychological adjustment to Long COVID symptoms, promote resilience, and facilitate coping, based on established psychotherapeutic techniques such as skills training, acceptance-based and identity-based principles.

The investigators will assess rates of recruitment, intervention engagement, and session attendance (feasibility), Veteran satisfaction (acceptability), treatment adherence (fidelity) and preliminarily explore response to Long COVID Coping and Recovery (LCCR). Findings will be used to make a final adaptation of the treatment materials and to develop a research protocol for a large scale RCT of LCCR for Veterans with Long COVID. This study will pilot test a well-specified, group-based intervention tailored to the unique needs of Veterans with Long COVID. The results of the proposed study will provide data to 1) identify adaptations needed to optimize LCCR for Veterans with Long COVID; 2) identify possible benefits of LCCR; 3) inform development of a large scale RCT of LCCR for Veterans with Long COVID.

DETAILED DESCRIPTION:
Epidemiological estimates suggest that approximately 11,390,400 Americans, and 90,300 Veterans in VA care experience symptoms for months after initial COVID-19 infection, a phenomenon known as Post-Acute COVID-19 Syndrome (PACS) or Long COVID. Common symptoms of Long COVID include prolonged fatigue, impairment of memory, concentration disorder, headache, pain, insomnia, anxiety, post-traumatic stress disorder (PTSD), and depression (Taquet et al., 2021). Longer term effects of COVID-19 have been reported in all age groups and demographics including persons with asymptomatic, mild, or severe initial COVID-19 infection. Despite Long COVID symptoms resulting in significant functional impairment, there are few empirically supported treatment approaches specifically designed to address this population. Many in the field contend that given the complexity and variability of Long COVID manifestations, successful treatment cannot be considered from a single organ point of view, but rather require a patient-tailored multidisciplinary approach that steps beyond amelioration of psychological symptoms (Ambrosino et al., 2021; Lerner et al., 2021). Long COVID treatment requires specialists across medical, neurological, rehabilitation, and mental health fields in conjunction with recovery-based approaches such as Whole Health, and Chaplain Services.

The investigator's proposed intervention, Long COVID Coping and Recovery (LCCR), aims to improve psychological adjustment to Long COVID symptoms, promote resiliency, and facilitate coping, all of which can impact functional status and quality of life. LCCR is designed to help to build a relevant and personally meaningful action plan to address the symptoms Veterans may be experiencing due to Long COVID and to assist Veterans with Long COVID in managing their illness, increasing function, and moving towards recovery. LCCR focuses on psychological adjustment and coping, and augments medical, rehabilitation, and neurological treatment for this population. The investigator's approach is based on the CHIME model of personal recovery which includes five overarching processes: 1) Connectedness; 2) Hope and optimism about the future; 3) Identity; 4) Meaning in life; and 5) Empowerment. The investigators will target the CHIME processes using established psychotherapeutic techniques such as skills training, acceptance-based and identity-based principles.

Based on adaptations from existing recovery-based and COVID-19 distress group interventions that the team has developed/piloted, the investigators have developed a treatment framework that consists of sixteen 60-minute weekly group sessions. The investigators specifically are designing a group intervention to build support and mitigate the loneliness associated with chronic conditions such as Long COVID The sessions will focus on the impact of Long COVID on mental and physical health, teach coping skills to foster resiliency and hope, and developing a sense of purpose and meaning in life even when living with a chronic condition like Long COVID.

Overall Goal: To pilot a Post-Acute COVID-19 Syndrome (PACS) psychotherapeutic intervention, "Long COVID Coping and Recovery" (LCCR) while collecting pilot data to assess its acceptability and feasibility.

Aim 1: Identify adaptations needed to optimize LCCR for Veterans with Long COVID through Veteran and stakeholder consultation.

Aim 2: Identify possible benefits of LCCR. Aim 3: Inform development of a large scale RCT of LCCR for Veterans with Long COVID.

ELIGIBILITY:
Inclusion Criteria:

1. U.S. Veteran
2. Ages 18-80
3. Positive screen for Long COVID (e.g. COVID-19 positive, diagnosed with a PCR test, an antibodies blood test, and or a diagnosis by a physician at the JJPVAMC Long COVID Clinic and symptoms lasting 1 month or longer after infection)
4. Participation in VA services at the JJPVAMC
5. Sufficient clinical stability and readiness to participate in group therapy as deemed by their VA service provider

Exclusion Criteria:

1. Active alcohol or opiate dependence requiring medically supervised withdrawal
2. Active psychosis
3. MINI Mental Status < 23 or inability to function in a group setting
4. Unable to operate telehealth platforms or other electronic devices
5. Non-English speaking
6. Lack of capacity to consent
7. Unable or unwilling to provide at least one contact for emergency purposes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S. Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant withdrew after signing the consent form before beginning treatment due to lack of interest in participating.
Period: Overall Study
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.363 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black/African American | 11
  Race: White/Caucasian | 5
  Race: Muti-racial | 2
  Race: Other | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) [Mean (Standard Deviation); unit: scores on a scale] — The Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm) contains 17 items that yield four scores. The worst scores for each item within Questions 1-10 form the symptom severity subscale (score 0-30), Questions 11-15 the functional disability subscale (0-15), Question 16 is the other symptoms subscale (score 0-25), and Question 17 is the overall health score (score 0-10). Higher scores indicate more severe symptoms, functional limitations, and perceived overall health. We used the symptom severity, functional disability, and overall health subscales.
  scores on a scale
    Functional disability | 8.05 (4.93)
    Symptom severity | 20.67 (4.63)
    Perceived overall health | 4.67 (1.98)
World Health Organization Disability Assessment Schedule, 2nd Version (WHODAS 2.0) [Mean (Standard Deviation); unit: scores on a scale] — The World Health Organization Disability Assessment Schedule 2.0 has 36 items ranging from 1 (None) to 5 (Extreme or cannot do). There are six domains: 1) understanding and communicating (scores 6-30), 2) getting around (scores 5-25), 3) self-care (scores 4-20), 4) getting along with people (scores 5-25), 5a) life activities-household (scores 4-20), 5b) life activities-school/work (scores 4-20), and 6) participation in society (scores 8-40). Items are summed for total scores. Higher scores indicate more difficulties due to health/mental health conditions. We used domains 1, 2, 3, 4, 5a, and 6.
  scores on a scale
    Domain 1 | 14.86 (5.11)
    Domain 2 | 14.71 (4.62)
    Domain 3 | 7.62 (2.73)
    Domain 4 | 10.71 (4.35)
    Domain 5 (Part A) | 11.71 (4.45)
    Domain 6 | 21.48 (8.87)
Suicidal Behaviors Questionnaire-Revised (SBQ-R) [Mean (Standard Deviation); unit: scores on a scale] — The Suicidal Behaviors Questionnaire-Revised (SBQ-R) is a four-item measure of suicide risk. Item 1 measures lifetime suicidal thoughts, plan, and attempt; item 2 measures the frequency of suicidal ideation over the past 12 months; item 3 measures the threat of suicide attempt; and item 4 measures the perceived likelihood of future suicidal behaviors. Items are recoded (item 1: 1-4; item 2: 1-5; item 3: 1-3; item 4: 0-6) and summed for total scores (3-18). Higher scores indicate more risk. Population: One participant was missing item 1 at baseline, so a total baseline SBQ-R could not be calculated.
  scores on a scale
    number analyzed (Participants) | 20
    (all) | 5.2 (3.14)
Measure of Current Status (MOCS - Part A) [Mean (Standard Deviation); unit: scores on a scale] — The Measure of Current Status (MOCS) has two parts (A and B). We used Part A, which consists of 13 items that measure participants' current self-perceived status on several skills. Item responses range from 0 (I cannot do this at all) to 4 (I can do this extremely well). We summed items for total scores (possible range: 0-52).
  scores on a scale | 26.19 (6.71)
Future Self-Continuity Questionnaire (FSCQ) [Mean (Standard Deviation); unit: scores on a scale] — The Future Self-Continuity Questionnaire (FSCQ) consists of 10 items on a 6-point metric measuring how individuals perceive themselves in the future in three areas: vividness of the future self, similarity with the future self, and positivity toward the future self. The total FSCQ score is averaged from all items and the total subscales scores are averaged from associated items (all total mean score range: 1-6). Higher subscale scores indicate increased levels of the domain, and higher total scores indicate increased future-self continuity. We used the total score and all subscale scores.
  scores on a scale
    Overall | 3.46 (1.00)
    Similarity subscale | 3.57 (1.46)
    Vividness subscale | 3.16 (0.79)
    Positivity subscale | 3.60 (1.53)
Patient Health Questionnaire-9 (PHQ-9) [Mean (Standard Deviation); unit: scores on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a 9-item questionnaire that assesses the presence and severity of depressive symptoms over the two weeks prior to completion. The items are assessed on a likert scale from 0 (not at all) to 3 (nearly every day). There is one additional item measuring how difficult the symptoms from items 1-9 have made daily life. Items 1-9 are summed for a total score (range from 0-27), with higher scores indicating increased depression severity.
  scores on a scale | 12.81 (6.38)
General Anxiety Disorder-7 (GAD-7) [Mean (Standard Deviation); unit: scores on a scale] — The Generalized Anxiety Disorder-7 (GAD-7) is a self-report measure based on DSM-IV GAD criteria that is used to screen for GAD and assess symptom severity. The scale has 7 items on a Likert scale from 0 (not at all) to 3 (nearly every day) asking about symptoms over the past two weeks. There is one additional item measuring how difficult the symptoms from items 1-7 have made daily life. Items 1-7 are summed for a total score (range 0-21), with higher scores indicating increased anxiety severity.
  scores on a scale | 10.87 (6.64)
Quality of Life Scale (QOLS) [Mean (Standard Deviation); unit: scores on a scale] — The Quality of Life Scale (QOLS) measures an individual's quality of life in five domains (i.e., material and physical well-being, relationships with other people, social, community, and civic activities, personal development and fulfillment, and recreation). Participants respond to each of 16 items using a scale of 1 (terrible) to 7 (delighted) to indicate levels of satisfaction among the domains. Items are summed for a total score (range: 16-112), with higher scores indicating greater quality of life.
  scores on a scale | 66.42 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Improvement Post-COVID-19 Over Time
Description: Our primary outcome will be changes in symptom severity and subsequent functional improvement (post-COVID-19), as measured by the Modified COVID-19 Yorkshire Rehabilitation Scale (C19-YRSm; Sivan et al., 2022). The C19-YRSm is a 17-item self-report scale adapted from the original 22-item COVID-19 Yorkshire Rehabilitation Scale (O'Connor et al., 2022). Items are rated on a scale from 0 (none of this symptom) to 3 (extremely severe level or impact). The C19-YRSm is divided into four subscales: symptom severity, functional disability, other symptoms (item 16), and overall health (item 17). The worst scores for each item within Questions 1-10 form the symptom severity subscale (score 0-30), Questions 11-15 the functional disability subscale (0-15), Question 16 is the other symptoms subscale (score 0-25), and Question 17 is the overall health score (score 0-10). Higher scores indicate more severity. We used the symptom severity, functional disability, and overall health subscales.
Time Frame: This outcome will be measured at 3 time points: Consent & baseline, immediately mid intervention (after the first 8 sessions), and immediately post intervention (after the second 8 sessions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  Functional disability - pre | 8.4 (4.78)
  Symptom severity - pre | 21.05 (4.39)
  Overall health - pre | 4.55 (1.96)
  Functional disability - post | 6.6 (3.2)
  Symptom severity - post | 17.25 (5.18)
  Overall health - post | 5.5 (1.7)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the functional disability subscale from pre- to post-intervention; Test type: Other; p = .06, paired t-test
Statistical Analysis 2: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the symptom severity subscale from pre- to post-intervention; Test type: Other; p = .004, paired t-test
Statistical Analysis 3: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the perceived overall health now subscale (1 item) from pre- to post-intervention; Test type: Other; p = .10, paired t-test

2. Secondary Outcome: Change in Health-Related Functional Status Over Time
Description: Changes in functional status as relates to health will be measured by the World Health Organization Disability Assessment Schedule, 2nd Version (WHODAS 2.0; Ustun et al., 2010). The WHODAS. 2.0 has 36 items ranging from 1 (None) to 5 (Extreme or cannot do). Items are summed for subscale scores. There are six domains: 1) understanding and communicating (scores 6-30), 2) getting around (scores 5-25), 3) self-care (scores 4-20), 4) getting along with people (scores 5-25), 5a) life activities-household (scores 4-20), 5b) life activities-school/work (scores 4-20), and 6) participation in society (scores 8-40). Higher scores indicate more difficulties due to health/mental health conditions in each domain. The WHODAS 2.0 has been validated in the general population and amongst those with non-acute health conditions and has a Cronbach's alpha of .96 (Saltychev et al., 2021). We used domains 1, 2, 3, 4, 5a, and 6.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  WHODAS 2.0 domain 1 - pre | 15.1 (5.12)
  WHODAS 2.0 domain 2 - pre | 15.1 (4.38)
  WHODAS 2.0 domain 3 - pre | 7.8 (2.67)
  WHODAS 2.0 domain 4 - pre | 10.95 (4.32)
  WHODAS 2.0 domain 5a - pre | 11.9 (4.48)
  WHODAS 2.0 domain 6 - pre | 22 (8.76)
  WHODAS 2.0 domain 1 - post | 14.15 (3.86)
  WHODAS 2.0 domain 2 - post | 14.05 (3.58)
  WHODAS 2.0 domain 3 - post | 7.25 (2.9)
  WHODAS 2.0 domain 4 - post | 11.2 (4.50)
  WHODAS 2.0 domain 5a - post | 10.9 (3.96)
  WHODAS 2.0 domain 6 - post | 20.35 (8.01)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 1 from pre- to post-intervention; Test type: Other; p = .46, paired t-test
Statistical Analysis 2: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 2 from pre- to post-intervention; Test type: Other; p = .20, paired t-test
Statistical Analysis 3: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 3 from pre- to post-intervention; Test type: Other; p = .42, paired t-test
Statistical Analysis 4: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 4 from pre- to post-intervention; Test type: Other; p = .84, paired t-test
Statistical Analysis 5: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 5 (part 1) from pre- to post-intervention; Test type: Other; p = .25, paired t-test
Statistical Analysis 6: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses domain 6 from pre- to post-intervention; Test type: Other; p = .26, paired t-test

3. Secondary Outcome: Change in Suicide Risk Over Time
Description: Changes in Suicide Risk will be measured by the Suicide Behaviors Questionnaire-Revised (SBQ-R; (Osman et al., 2001). The SBQ-R is a four-item measure of suicide risk. Item 1 measures lifetime suicidal thoughts, plan, and attempt; item 2 measures the frequency of suicidal ideation over the past 12 months; item 3 measures the threat of suicide attempt; and item 4 measures the perceived likelihood of future suicidal behaviors. Items are recoded (item 1: 1-4; item 2: 1-5; item 3: 1-3; item 4: 0-6) and summed for total scores (3-18). Higher scores indicate more risk.
Time Frame: as for outcome 1
Population: One participant was missing item 1 of the SBQ-R and was not included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 19
score on a scale
  SBQ-R - pre | 4.89 (2.9)
  SBQ-R - post | 5.05 (3.22)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the SBQ-R total score from pre- to post-intervention; Test type: Other; p = .89, Wilcoxon test

4. Secondary Outcome: Change in Self-perceived Status on Several Skills Over Time
Description: The Measure of Current Status (MOCS) has two parts (A and B). We used Part A, which consists of 13 items that measure participants' self-perceived proficiency in skills necessary for responding to challenges of everyday life. Item responses range from 0 (I cannot do this at all) to 4 (I can do this extremely well). We summed items for total scores (possible range: 0-52). Higher scores indicate greater self-perceived proficiency of the skills listed. Reliability alphas range from 0.71 to 0.89 (Antoni et al., 2006).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  MOCS - pre | 27.05 (5.58)
  MOCS - post | 27.50 (6.12)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the MOCS (part A) from pre- to post-intervention; Test type: Other; p = .80, paired t-test

5. Secondary Outcome: Change in Identity Concerns Over Time
Description: Changes in identity concerns will be assessed with the Future Self-Continuity Questionnaire (FSCQ). The FSCQ measures how individuals perceive themselves in the future in three areas: vividness of the future self, similarity with the future self, and positivity toward the future self. Items range from 1-6. The total FSCQ score is averaged from all items and the total subscales scores (vividness, similarity, and positivity) are averaged from associated items (all total mean scores range from 1-6). Higher subscale scores indicate increased levels of the domain, and higher total scores indicate increased future-self continuity. The FSCQ has demonstrated high levels of reliability ( =.85) and validity. We used the total score and all three subscale scores.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  FSCQ total score - pre | 3.52 (.99)
  FSCQ similarity subscale - pre | 3.68 (1.42)
  FSCQ vividness subscale - pre | 3.18 (.8)
  FSCQ positive subscale - pre | 3.65 (1.55)
  FSCQ total score - post | 3.54 (1.03)
  FSCQ similarity subscale - post | 3.5 (1.34)
  FSCQ vividness subscale - post | 3.27 (.93)
  FSCQ positive subscale - post | 3.87 (1.22)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the FSCQ score (all items) from pre- to post-intervention; Test type: Other; p = .92, paired t-test
Statistical Analysis 2: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the FSCQ similarity subscale from pre- to post-intervention; Test type: Other; p = .90, Wilcoxon test (paired)
Statistical Analysis 3: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the FSCQ vividness subscale from pre- to post-intervention; Test type: Other; p = .74, paired t-test
Statistical Analysis 4: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the FSCQ positivity subscale from pre- to post-intervention; Test type: Other; p = .44, paired t-test

6. Secondary Outcome: Change in Depression Over Time
Description: Changes in depressive symptoms will be measured with the Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001). The PHQ-9 is a 9-item depression module from the full PHQ with each item representing a depressive symptom. Items are scored on a scale ranging from 0 (not at all) to 3 (nearly every day) to assess the frequency of each symptom over a two-week period. Items are summed for a total score (range from 0-27), with higher scores indicating increased depression severity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  PHQ-9 - pre | 12.95 (6.52)
  PHQ-9 - post | 8.65 (4.90)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the PHQ-9 from pre- to post-intervention; Test type: Other; p = .003, paired t-test

7. Secondary Outcome: Change in Anxiety Over Time
Description: Changes in anxiety symptoms will be measured with the GAD-7 Anxiety (Spitzer et al., 2006). The GAD-7 is a brief self-report measure to assess symptomatology and severity related to Generalized Anxiety Disorder over the course of the last two weeks. The scale has 7 items with a 4-point Likert scale responses (0 = Never to 3 = almost every day). Items are summed for a total score (ranging from 0 to 21), with higher scores indicating increased anxiety severity. The GAD-7 has excellent reliability and validity (Spitzer et al., 2006).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  GAD-7 - pre | 11.01 (6.78)
  GAD-7 - post | 7.95 (5.56)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the GAD-7 from pre- to post-intervention; Test type: Other; p = .01, paired t-test

8. Secondary Outcome: Change in Quality of Life Over Time
Description: Changes in quality of life will be measured with the The Quality of Life Scale (QOLS; Burckhardt & Anderson, 2003). The QOLS measures quality of life relevant to diverse patient groups with chronic illness across 6 domains: material and physical well-being, relationships with other people, social, community, and civic activities, personal development and recreation, and independence. There are 16 items with a response scale ranging from 1 (terrible) to 7 (delighted) to indicate levels of satisfaction among the domains. Items are summed for a total score (range: 16-112), with higher scores indicating greater quality of life.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  QOLS - pre | 66.34 (15.69)
  QOLS - post | 72.75 (14.09)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; This analysis uses the QOLS from pre- to post-intervention; Test type: Other; p = .04, paired t-test

9. Secondary Outcome: Changes in Intervention Acceptability, Feasibility, and Appropriateness Over Time.
Description: Changes in Intervention Acceptability, Feasibility, and Appropriateness will be measured by Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) (Weiner et al., 2017) at each assessment point. These measures are considered "leading indicators" of implementation success (acceptability and feasibility of intervention and intervention appropriateness) (Proctor et al., 2011). Each measure has four items rated from 1 (completely disagree) to 5 (completely agree). Items are averaged for total scores, and higher scores indicate higher acceptability (AIM), appropriateness (IAM), and feasibility (FIM).
Time Frame: This outcome will be measured at 2 time points: Consent & baseline and immediately post intervention (after the second 8 sessions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
Number analyzed (Participants) | 20
score on a scale
  Acceptability - pre | 4.04 (.80)
  Appropriateness - pre | 4.16 (.77)
  Feasibility - pre | 3.96 (.70)
  Acceptability - post | 4.26 (.75)
  Appropriateness - post | 4.20 (.79)
  Feasibility - post | 4.15 (.75)
Statistical Analysis 1: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; Test type: Other — The AIM measures an intervention's acceptability. Therefore, the goal is not change over time, the goal is to assess, descriptively, post-intervention acceptability. Because we assessed this measure at baseline (with "expectations of the future treatment"), we provide a paired t-test with the AIM at pre- and post-intervention; p = .24, Paired t-test
Statistical Analysis 2: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; Test type: Other — The IAM measures an intervention's appropriateness. Therefore, the goal is not change over time, the goal is to assess, descriptively, post-intervention appropriateness. Because we assessed this measure at baseline (with "expectations of the future treatment"), we provide a paired t-test with the IAM at pre- and post-intervention; p = .82, Paired t-test
Statistical Analysis 3: Comparison: Long COVID Coping and Recovery (LCCR) Intervention; The FIM measures an intervention's feasibility. Therefore, the goal is not change over time, the goal is to assess, descriptively, post-intervention feasibility. Because we assessed this measure at baseline (with "expectations of the future treatment"), we provide a paired t-test with the FIM at pre- and post-intervention; Test type: Other; p = .38, Paired t-test

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the course of participant enrollment in the study (about 13 months).
Arm/Group | Long COVID Coping and Recovery (LCCR) Intervention
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 9/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long COVID Coping and Recovery (LCCR) Intervention (N=21)
Abdominal Surgery (Surgical and medical procedures) | 1 (1)
Gynecological Surgery (Reproductive system and breast disorders) | 1 (1)
Emergency Department visit for chest pain (Cardiac disorders) | 1 (1)
Emergency Department visit and hospitalization for dizziness and chest pain (Cardiac disorders) | 1 (1)
Emergency Department visit and hospitalization for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac Surgery (Cardiac disorders) | 1 (1)
Emergency Department visit and hospitalization for COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hip Replacement Surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Long COVID Coping and Recovery (LCCR) Intervention (N=21)
Emergency Department visit for cough and fever (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emergency Department visit for COVID-19 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Oral Surgery (Surgical and medical procedures) | 1 (1)
Emergency Department visit for shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hand Surgery (Surgical and medical procedures) | 1 (1)
Emergency Department visit for back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Emergency Department visit for hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Emergency Department visit for EKG irregularity (Cardiac disorders) | 1 (1)
Emergency Department visit for groin pain and hyperglycemia (Endocrine disorders) | 1/1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05453201/Prot_001.pdf
  • Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05453201/SAP_002.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT05453201/ICF_000.pdf